CLINICAL TRIAL: NCT02054884
Title: Phase II Study of the Tumor-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Paclitaxel in Patients With Metastatic Merkel Cell Carcinoma
Brief Title: F16IL2 Plus Paclitaxel in Metastatic Merkel Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2TAXO-03/12
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Merkel Cell Carcinoma
Keywords: Interleukin, IL2, F16, monoclonal, antibody, cytokine Paclitaxel, Merkel cell carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: F16IL2 in combination with paclitaxel (Experimental)
  Interventions: Drug: Arm A: F16IL2 in combination with paclitaxel
- Arm B: Paclitaxel (Experimental)
  Interventions: Drug: Arm B: Paclitaxel

INTERVENTIONS:
Drug: Arm A: F16IL2 in combination with paclitaxel — Intravenous (i.v.) 1 hour infusions of paclitaxel 90 mg/m^2 followed, after 30 min pause, by 3 hour i.v. infusions of F16IL2 35 Mio IU on days 1, 8, 15 of each 28 day cycle.
  Patients will receive 4 week cycles of study therapy for a maximum of 24 weeks, or until disease progression, unacceptable toxicity or withdrawal of consent.
  Arms: Arm A: F16IL2 in combination with paclitaxel
Drug: Arm B: Paclitaxel — Intravenous (i.v.) 1 hour infusions of Paclitaxel 90 mg/m^2 on days 1, 8, 15 of each 28 day cycle.
  Patients will receive 4 week cycles of study therapy for a maximum of 24 weeks, or until disease progression, unacceptable toxicity or withdrawal of consent.
  Arms: Arm B: Paclitaxel

SUMMARY:
There is no standard treatment for Merkel cell carcinoma(MCC), as no randomized trials have been conducted to establish standard of care. Despite a sizable number of objective responses induced by combination cyototoxic chemotherapy, a prolongation of patients overall survival has never been demonstrated.

This open-label, randomized, double-arm, multi-centre, phase II study of F16IL2 in combination with paclitaxel versus paclitaxel monotherapy, proposes to test the therapeutic efficacy of F16IL2 plus paclitaxel in patients with metastatic Merkel cell carcinoma, who are not amenable to surgery.

A total of 90 patients with Merkel cell carcinoma will be enrolled and treated during the study; 45 patients will receive the combination treatment of F16IL2 and paclitaxel (Arm A), and 45 patients will receive paclitaxel monotherapy (Arm B).

DETAILED DESCRIPTION:
F16IL2 has been studied in two clinical pase I/II trials in patients with different advanced cancer types. One of them (Nr. EudraCT: 2007-006457-42) tested the administration of therapeutic doses of paclitaxel (up to 90 mg/m2 on a weekly basis) together with escalating doses of F16IL2 (from 5 Mio IU of IL2 equivalents in a weekly administration schedule, until definition of MTD). More than 40 patients were treated in this clinical trial. As of today, the highest F16IL2 dose tested corresponds to 45 Mio IU, but the dose escalataion of the F16IL2/paclitaxel combination study is still ongoing.

In general, treatment of patients with F16IL2 plus paclitaxel was very well tolerated not exceeding the expected toxicity of chemotherapy alone. Multiple objective and durable tumor responses were observed in the F16IL2/paclitaxel combination trial(particularly in patients with non small cell lung cancer or melanoma who had previously failed several lines of chemotherapy). In addition to several disease stabilizations of previously progressive patients.

Paclitaxel promotes the assembly of microtubules from tubulin dimers and stabilizes microtubules by preventing depolymerisation. This stability results in the inhibition of the normal reorganization of the microtubule network that is essential for vital interphase and mitotic cellular functions. In addition, paclitaxel reduces abnormal arrays or bundles of microtubules throughout the cell cycle and multiple asters of microtubules during mitosis.

F16 is a human recombinant antibody fragment in the scFv (single chain Fragment variable) format that is directed against tenascin C, an angiogenesis marker common to most solid tumors independent of the tumor type. ScFv(F16) selectively localizes in tumor tissues in animal models as demonstrated both histologically and during mechanistic studies involving mice transfected with orthotopic human tumours.

IL2, the human cytokine interleukin-2, is a potent stimulator of the immune response. It has a central role in the regulation of T cell responses and effects on other immune cells such as natural killer cells, B cells, monocyte/macrophages and neutrophils (Smith, 1988). IL2 can induce tumor regression through its ability to stimulate a potent cell-mediated immune response in vivo (Rosenberg, 2000).

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic Merkel cell carcinoma (MCC) not amenable to surgery and who have not received previous systemic therapy with taxanes; diagnosis of MCC must be histologically confirmed (evaluation of primary lesions or advanced disease) and endorsed by the IMMOMEC central dermatopathology center (central review of diagnosis at the Department of General Dermatology, Medical University of Graz). Patients must be amenable for paclitaxel treatment according to the discretion of the principal investigator
* Patients aged ≥ 18 ≤ 75 years
* ECOG performance status ≤ 1
* Patients must have measurable disease including cutaneous and subcutaneous metastases as defined by RECIST v.1.1 criteria or immune related response Criteria (irRC) as assessed by CT or MRI and/or ultrasound within 4 weeks before the first study drug administration.
* All acute side effects from any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) Grade ≤ 1;.
* Adequate hematologic, liver and renal function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, haemoglobin (Hb) ≥ 9.0 g/dl
  * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and/or aspartate aminotransferase ≤ 3 x upper limit of reference range (ULN), and total bilirubin ≤ 2.0 mg/gL unless liver involvement by the tumor, in which case the transaminase levels could be ≤ 5 x ULN
  * Creatinine ≤ 1.5 UL or 24 h creatinine clearance ≥ 50 mL/min
* Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment
* If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug
* Evidence of a personally signed and dated EC-approved Informed Consent form indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Life expectancy of less than 3 months
* Any previous taxanes therapy
* Previous or concurrent CLL patients
* Any other malignancy from which the patient has been disease-free for less than 2 years prior to study entry, with the exception of adequately treated and cured cervical carcinoma in situ, basal or squamous cell carcinoma, superficial bladder cancer, or in situ melanoma
* Presence of uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study
* Presence of known brain metastases
* Chronic-active hepatitis B, C, or HIV
* Severe cardiovascular disease:

  * History of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris
  * Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria)
  * Irreversible cardiac arrhythmias requiring permanent medication
  * LVEF < 50% and/or abnormalities observed during baseline 2D-ECHO or 12-lead ECG investigations
  * Uncontrolled hypertension
  * Ischemic peripheral vascular disease (Grade IIb-IV)
* Severe rheumatoid arthritis; or other uncontrolled autoimmune disease
* Severe diabetic retinopathy
* History of allograft or stem cell transplantation
* Major trauma including major surgery (e.g. visceral surgery) within 4 weeks of administration of study treatment
* Known history of allergy to IL-2, taxanes, cremophor or other intravenously administered human proteins/peptides/antibodies
* Pregnancy or breast-feeding. Female patient must agree to use effective contraception, or be surgically sterile or postmenopausal. The definition of effective contraception will be based on the European guideline ICH M3 rev 2.
* Treatment with an investigational study drug within four weeks before beginning of treatment with F16IL2
* Previous treatment with monoclonal antibodies for biological therapy in the four weeks before administration of study treatment
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of F16IL2 in combination with paclitaxel vs. paclitaxel monotherapy (RECIST v1.1, irRC) | 12 months

SECONDARY OUTCOMES:
Overall survival rate | 12 months
Treatment efficacy (ORR, DCR) | 36 months
Safety and tolerability of the combination treatment with F16IL2 and paclitaxel | 36 months
  Evaluation of the type and the number of adverse events eventually present

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen C. Becker, Prof., Principal Investigator — Medical University of Graz, Austria
Locations (8):
- Medical University Hospital, Graz, Austria
- Herlev- University Hospital, Herlev, Denmark
- Saint-Louis- Hospital, Paris, France
- Germany (3):
  - Charité- Medical University Hospital, Berlin
  - Universitätsklinik Essen, Essen
  - Eberhard-Karls- University Hospital, Tübingen
- ICMiD- University Hospital, Barcelona, Spain
- Nottingham Trent- University Hospital, Nottingham, United Kingdom